CLINICAL TRIAL: NCT01227850
Title: Leptin and IGF1; Diagnostic Markers of Refeeding Syndrome and Mortality
Brief Title: Leptin, IGF1 and the Refeeding Index
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Carel Le Roux, King's College Hospital
Other Study IDs: Refeedingindex0810
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Refeeding Syndrome
Keywords: Leptin; IGF1; Refeeding Index; Hypophosphataemia; Primary focus of the study was to detemine whether the 'Refeeding Index', could reliably predict,that the refeeding syndrome would occur
MeSH Terms: conditions — Refeeding Syndrome; Hypophosphatemia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parenteral nutrition patients.

SUMMARY:
Background and study hypothesis:

Refeeding syndrome is a dangerous condition which could arise if patients who have had little or no food for many days, are started on any form of feeding. The metabolic consequences of this condition could affect the heart, lungs and nervous system of the patient and cause serious imbalance in the level of salts in the body.

The available guidelines for predicting that refeeding syndrome may occur are very subjective since they depend mainly on a history which is sometimes difficult to obtain from the patient.

The main biochemical landmark that refeeding syndrome has occurred is a fall in the phosphate levels once feeding has been started. There are currently no biochemical markers that can identify patients at risk of developing refeeding syndrome.

Leptin and IGF1 are hormones which have been observed to go down if someone has had little or no food for a while. The investigators therefore hypothesized that using a combination of leptin and IGF1 values in a 'Refeeding Index' would make the latter a useful biochemical marker to predict that refeeding may occur, hence take the precautionary measures to avoid its occurrence before starting feeding.

Design: Thirty five consecutive patients referred for commencement of parenteral nutrition (PN) were included. Serum leptin and IGF1 were measured prior to starting PN. Electrolytes, liver and renal function tests were measured before and daily for one week after initiating PN. The primary outcome was a decrease in phosphate on day two or three after initiating PN. A 'Refeeding Index' (RI) was defined as leptin x IGF1 divided by 2800 to produce a ratio of 1.0 in patients who are well nourished.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred for parenteral nutrition at King's College Hospital between January and April 2009.

Exclusion Criteria:

* Non adult patients (less than 18 years of age).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to our department at King's College Hospital, for commencement of parenteral nutrition (PN).These included all ages above 18 and both sexes. Consent to commence PN was taken from the patients prior to starting it. Daily bloods were taken for routine laboratory analysis as part of the usual patient care.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel W Le Roux, MRCPath, MRCP, PhD, Principal Investigator — King's College Hospital NHS Trust

REFERENCES:
- [Derived] Goyale A, Ashley SL, Taylor DR, Elnenaei MO, Alaghband-Zadeh J, Sherwood RA, le Roux CW, Vincent RP. Predicting refeeding hypophosphataemia: insulin growth factor 1 (IGF-1) as a diagnostic biochemical marker for clinical practice. Ann Clin Biochem. 2015 Jan;52(Pt 1):82-7. doi: 10.1177/0004563214523739. Epub 2014 Mar 7. PMID 24609720